CLINICAL TRIAL: NCT05219669
Title: An Open-Label, Three-Period, Three-Treatment, Six-Sequence, Randomized Crossover Study of the Pharmacokinetics of Intranasal Nalmefene in Healthy Volunteers Using Three Dosing Regimens
Brief Title: Pharmacokinetic Evaluation of Intranasal Nalmefene Using Three Dosing Regimens
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Opiant Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OPNT003-PK-002
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Results first posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-02

CONDITIONS: Opioid Overdose
Keywords: Pharmacokinetics
MeSH Terms: conditions — Opiate Overdose | interventions — nalmefene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intranasal Nalmefene 1 Spray in 1 Nostril (Experimental): 3 mg IN Nalmefene Hydrochloride dose (one 0.1 mL spray of a 30 mg/mL solution in one nostril)
  Interventions: Drug: Nalmefene Hydrochloride
- Intranasal Nalmefene 2 Sprays in 1 Nostril (Experimental): 6 mg IN Nalmefene Hydrochloride dose (two 0.1 mL sprays of a 30 mg/mL solution in one nostril)
  Interventions: Drug: Nalmefene Hydrochloride
- Intranasal Nalmefene 1 Spray in Each Nostril (Experimental): 6 mg IN Nalmefene Hydrochloride dose (one 0.1 mL spray of a 30 mg/mL solution in each nostril)
  Interventions: Drug: Nalmefene Hydrochloride

INTERVENTIONS:
Drug: Nalmefene Hydrochloride — 30 mg/mL solution

SUMMARY:
This study is to compare the pharmacokinetics (how the body absorbs, breaks down and eliminates drug from your body) of nalmefene when given as a single dose intranasally (IN;into the nose), as a single dose in each nostril and as two doses in one nostrils; and to evaluate the safety and tolerability of nalmefene IN.

DETAILED DESCRIPTION:
Open-label, randomized, 3-period, 3-treatment, 6-sequence, ranodmised crossover study in 24 healthy volunteers. Subjects will be assigned to each of the 6 possible sequences. Each subject will receive 3 intranasal (IN) nalmefene doses:

* 3mg IN dose (one 0.1mL spray of a 30mg/mL solution in one nostril)
* 6mg IN dose (one 0.1mL spray of a 30mg/mL solution in each nostril)
* 6mg IN dose (two 0.1mL sprays of a 30mg/mL solution in one nostril)

There will be a 6 day washout period between doses. Screening can occur up to 28 days before admission, subjects will then stay in the inpatient facility for 16 days to complete the treatment phase of the study and will be discharged following completion of the discharge procedures at the end of the last period. Subjects will be called 3 to 5 days after discharge to inquire concerning Adverse Events (AEs) and concomitant medications since discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 55 years inclusive
* BMI ranging from 18 to 30 kg/m2, inclusive
* Adequate venous access
* Subjects must be non-smokers
* On screening and admission, the following standards had to be met before dosing and were permitted to be repeated once:

  * Systolic blood pressure: 140 mmHg or less and equal to or greater than 90 mmHg
  * Diastolic blood pressure: 90 mmHg or less and equal to or greater than 55 mmHg
  * Heart rate: 100 beats per minute (bpm) or less and equal to or greater than 40 bpm
  * Respiratory rate: 20 respirations per minute (rpm) or less and equal to or greater than 8 rpm

Exclusion Criteria:

* History of clinically significant disease
* Significant trauma injury, major surgery, open biopsy within 30 days prior to screening
* Following an abnormal diet 4 weeks prior to screening
* Use of prescribed or over the counter medications, dietary supplements, herbal products, vitamins or opioid analgesics 14 days before intervention and throughout the study
* Use of enzyme altering drugs 30 days before intervention or during the study
* Use of nasal products 28 days before intervention and throughout the study
* Experimental agents used at least 8 weeks prior to initial dosing for a period equivalent to 5 half-lives of the agent (whichever was longer).
* Positive urine drug test for alcohol, opioids, cocaine, methamphetamine, benzodiazepines, tetrahydrocannabinol (THC), barbiturates, or methadone at screening or admission.
* Previous or current opioid, alcohol, or other drug dependence (excluding nicotine and caffeine)
* Positive urine screen for cotinine (smoking and the use of tobacco products were not permitted for 4 weeks prior to the first dose of study drug and throughout the duration of the study).
* An ECG QTcF interval >450 msec for males and > or equal to 470 msec for females.
* Clinically significant concurrent medical conditions
* Donated or received blood 30 days before intervention
* Women who are pregnant or breastfeeding at screening and prior to each administration of study drug
* Women of childbearing potential unless surgically sterile or use effective contraception
* Male subjects of childbearing potential that do not agree to use effective contraception
* Male subjects who plan to donate sperm or have female partner(s) who are pregnant, lactating or planning to attempt to become pregnant during the study or within 4 weeks after completion of the study
* Positive test for HBsAg, HCVAb, or HIVAb at screening
* Current or recent upper respiratory tract infection
* Current or recent use of any decongestants
* Allergic to nalmefene
* Those who would not abstain from engaging in strenuous exercise during the inpatient stay of the study.
* Those who would not abstain from consuming poppy seed or similar opium derived food stuff during the study.
* Those who would not abstain from ingesting alcohol, drinks containing xanthine >500 mg/day (e.g., Coca Cola®, coffee, tea, etc.), or grapefruit/grapefruit juice 72 hours before initial dosing and throughout the duration of the study.
* Those deemed unlikely to be able to comply with the requirements of the protocol.
* Those with any laboratory tests from samples taken at screening considered clinically significant.
* Those with a known intolerance to continuous ECG lead adhesive exposure.
* Brief Smell Identification Test (BSIT) score < 5 at screening.
* Those with a known hypersensitivity reaction to plastic.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ingela Danielsson, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- WorldWide Clinical Trials, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crystal R, Ellison M, Purdon C, Skolnick P. Pharmacokinetic Properties of an FDA-approved Intranasal Nalmefene Formulation for the Treatment of Opioid Overdose. Clin Pharmacol Drug Dev. 2024 Jan;13(1):58-69. doi: 10.1002/cpdd.1312. Epub 2023 Jul 27. PMID 37496452

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: "Sequence 1" represents subjects taking
  * Treatment "A" in period 1 (3 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in one nostril])
  * Treatment "B" in period 2 (6 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in each nostril])
  * Treatment "C" in period 3 (6 mg IN nalmefene dose [two 0.1 mL sprays of a 30 mg/mL solution in one nostril])
- Sequence 2: "Sequence 2" represents subjects taking
  * Treatment "B" in period 1 (6 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in each nostril])
  * Treatment "C" in period 2 (6 mg IN nalmefene dose [two 0.1 mL sprays of a 30 mg/mL solution in one nostril])
  * Treatment "A" in period 3 (3 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in one nostril])
- Sequence 3: "Sequence 3" represents subjects taking
  * Treatment "C" in period 1 (6 mg IN nalmefene dose [two 0.1 mL sprays of a 30 mg/mL solution in one nostril])
  * Treatment "A" in period 2 (3 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in one nostril])
  * Treatment "B" in period 3 (6 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in each nostril])
- Sequence 4: "Sequence 4" represents subjects taking
  * Treatment "A" in period 1 (3 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in one nostril])
  * Treatment "C" in period 2 (6 mg IN nalmefene dose [two 0.1 mL sprays of a 30 mg/mL solution in one nostril])
  * Treatment "B" in period 3 (6 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in each nostril])
- Sequence 5: "Sequence 5" represents subjects taking
  * Treatment "B" in period 1 (6 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in each nostril])
  * Treatment "A" in period 2 (3 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in one nostril])
  * Treatment "C" in period 3 (6 mg IN nalmefene dose [two 0.1 mL sprays of a 30 mg/mL solution in one nostril])
- Sequence 6: "Sequence 6" represents subjects taking
  * Treatment "C" in period 1 (6 mg IN nalmefene dose [two 0.1 mL sprays of a 30 mg/mL solution in one nostril])
  * Treatment "B" in period 2 (6 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in each nostril])
  * Treatment "A" in period 3 (3 mg IN nalmefene dose [one 0.1 mL spray of a 30 mg/mL solution in one nostril])
Period: Period 1 (1 Day)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 (Crossover study 24 subjects started the study. 1 subject did not complete this leg.) | 4 (Crossover study 24 subjects started the study.) | 4 (Crossover study 24 subjects started the study. 1 subject did not complete this leg.) | 4 | 4 | 4
Completed | 4 | 4 | 3 (1 subject withdrew consent at Period 1 prior to the second period.) | 4 | 4 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Washout (6 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 3 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (1 Day)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 3 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (6 Days)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 3 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (1 Day)
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 4 | 4 | 3 | 4 | 4 | 4
Completed | 4 | 4 | 3 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6 | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (5.91) | 32.0 (9.20) | 35.0 (8.29) | 37.5 (12.40) | 28.0 (6.73) | 27.0 (6.06) | 31.2 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 1 | 3 | 3 | 15
  Male | 2 | 1 | 1 | 3 | 1 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 0 | 1 | 3 | 2 | 10
  White | 2 | 2 | 3 | 2 | 1 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 4 | 4 | 4 | 24
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.28 (4.853) | 25.80 (2.226) | 24.30 (2.426) | 23.18 (4.921) | 23.00 (2.362) | 24.58 (3.222) | 24.52 (3.357)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Maximum concentration of plasma nalmefene comparing 1 dose of IN in one nostril to 2 doses of IN in 1 nostril to 1 dose of IN in each nostril
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Intranasal Nalmefene 1 Spray in 1 Nostril | Intranasal Nalmefene 2 Sprays in 1 Nostril | Intranasal Nalmefene 1 Spray in Each Nostril
Number analyzed (Participants) | 23 | 24 | 23
ng/ml | 10.8 (4.87) | 18.9 (11.2) | 22.2 (13.5)

2. Primary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time to maximum concentration of plasma nalmefene comparing 1 dose of IN in one nostril to 2 doses of IN in 1 nostril to 1 dose of IN in each nostril
Time Frame: 48 hours
Measure: Median (Full Range); unit: hours
Arm/Group | Intranasal Nalmefene 1 Spray in 1 Nostril | Intranasal Nalmefene 2 Sprays in 1 Nostril | Intranasal Nalmefene 1 Spray in Each Nostril
Number analyzed (Participants) | 23 | 24 | 23
hours | 0.267 [0.167 to 2.03] | 0.25 [0.117 to 3] | 0.25 [0.117 to 2.03]

3. Primary Outcome: Area Under the Curve (AUC)
Description: Area under the curve of plasma nalmefene comparing 1 dose of IN in one nostril to 2 doses of IN in 1 nostril to 1 dose of IN in each nostril
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: AUCinf (ng·h/mL)
Arm/Group | Intranasal Nalmefene 1 Spray in 1 Nostril | Intranasal Nalmefene 2 Sprays in 1 Nostril | Intranasal Nalmefene 1 Spray in Each Nostril
Number analyzed (Participants) | 23 | 24 | 23
AUCinf (ng·h/mL) | 46.8 (10.1) | 85.7 (18.7) | 89.5 (17.0)

4. Primary Outcome: Half-life (t1/2)
Description: Half life of plasma nalmefene comparing 1 dose of IN in one nostril to 2 doses of IN in 1 nostril to 1 dose of IN in each nostril
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Intranasal Nalmefene 1 Spray in 1 Nostril | Intranasal Nalmefene 2 Sprays in 1 Nostril | Intranasal Nalmefene 1 Spray in Each Nostril
Number analyzed (Participants) | 23 | 24 | 23
hour | 11.4 (2.51) | 11.3 (1.86) | 11.3 (1.87)

ADVERSE EVENTS:
Time Frame: Subjects were collected AE from baseline to day 15 with a +3 to 5 day follow-up. During the 15 days in clinic they received one of the three doing regimens on day 1, 7 and 13.
Arm/Group | Intranasal Nalmefene 1 Spray in 1 Nostril | Intranasal Nalmefene 2 Sprays in 1 Nostril | Intranasal Nalmefene 1 Spray in Each Nostril
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 9/23 | 16/24 | 12/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Nalmefene 1 Spray in 1 Nostril (N=23) | Intranasal Nalmefene 2 Sprays in 1 Nostril (N=24) | Intranasal Nalmefene 1 Spray in Each Nostril (N=23)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3
Nausea (Gastrointestinal disorders) | 1 | 1 | 5
Headache (Nervous system disorders) | 3 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT05219669/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/69/NCT05219669/SAP_001.pdf